CLINICAL TRIAL: NCT04853680
Title: A Prospective Randomized Controlled Study of Whether Anti-adhesion Barrier Can Prevent Voice Quality After Thyroidectomy.
Brief Title: Effect of Anti-adhesion Barrier on the Voice Quality After Thyroidectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Jin Wook Yi, Assistant Professor, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-12-023-001
Record Dates: First submitted 2021-04-11; First posted 2021-04-21 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Thyroid Nodule; Thyroid Cancer; Voice Disorders
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms; Voice Disorders

STUDY DESIGN:
Intervention Model Description: Treatment: Use of Anti-adhesion barrier on the thyroidectomy space Control: No use of anti-adhesion barrier
Who Masked: Participant
Masking Description: Participants do not know about the use of anti-adhesion agents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Use of Anti-adhesion barrier on the thyroidectomy space. After the thyroidectomy, anti-adhesion barrier will be applied on the thyroidectomy space, around the trachea, cricothyroid muscle and platysma muscle before the closure of surgical wound.
  Interventions: Device: Anti-adhesion barrier (Collarbarrier)
- Control (No Intervention): No use of anti-adhesion barrier. After the thyroidectomy, don't use the anti-adhesion barrier before the wound closure.

INTERVENTIONS:
Device: Anti-adhesion barrier (Collarbarrier) — Collagen derived anti-adhesion barrier
  Arms: Treatment

SUMMARY:
To determine whether the use of anti-adhesion barrier after thyroid surgery can prevent the voice changes after surgery, using objective voice-related indicators.

DETAILED DESCRIPTION:
* Randomized controlled study
* Including 40 patients in each arm
* Treatment: anti-adhesion barrier apply on the thyroidectomy space
* Control: No use of anti-adhesion barrier
* Primary outcome: VHI-30 (Voice handicap index)
* Secondary outcome: findings from stroboscopy, CSL (Computerize Speech Lab)
* Outcome measurement: preoperative, post-operative 3 months, post-operative 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open thyroidectomy for thyroid cancer
* Patients whose tumor size is less than 4cm
* Patients who are not suspected of surrounding organ involvement (T4) or metastasis to central lymph nodes in preoperative imaging
* Patients with no history of voice-related diseases prior to surgery
* Patients with normal movement of both vocal cords in the preoperative vocal cord examination
* Patients who consented to the study and obtained consent for the study

Exclusion Criteria:

* Patients with uncontrolled high blood pressure, diabetes, chronic renal failure, coagulation disease, etc.
* History of cardiovascular disease (angina pectoris, heart failure, myocardial infarction, cerebral infarction, cerebral hemorrhage, etc.)
* Medical history of drug or substance disorder (alcohol, etc.)
* Patients with diseases related to airways, esophagus, and vocal cords (vocal palsy, vocal cord polyps, etc.)
* Patients who have already had adhesions in the foreground due to radiation therapy or surgery on the foreground in the past.
* Patients with a history of keloid or hypertrophic scars
* Patients planning to perform lateral cervical lymph node dissection
* Patients with medical thyroid disease, such as Graves' disease and thyroid inflammation in need of treatment
* Pregnant or lactating female patients
* Other patients who are in charge of clinical trials as unsuitable for participation in the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Voice Handicap Index - 30 (VHI-30) | Preoperative 1 day
  Overall score of VHI (Total 30 points)
Voice Handicap Index - 30 (VHI-30) | Postoperative 3 months
  Overall score of VHI (Total 30 points)
Voice Handicap Index - 30 (VHI-30) | Postoperative 9 months
  Overall score of VHI (Total 30 points)

SECONDARY OUTCOMES:
Voice range profile (VRP) | Preoperative 1 day, Post-operative 3 months, Post-operative 9 months.
  Mininum Hz, Maximal Hz
GRBAS score | Preoperative 1 day, Post-operative 3 months, Post-operative 9 months.
  Grade, Rough, Breathy, Asthenic, Strained score. (0-3 points in each parameter)

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No
In order to protect the privacy of patients, the original data of the study will not be disclosed.